CLINICAL TRIAL: NCT00457769
Title: Phase 1 Study of Aricept Plus a Behavioral Strategy to Improve Functional Tasks in Vascular Dementia
Brief Title: Aricept to Improve Functional Tasks in Vascular Dementia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, A. M. Barrett, MD, Director, Stroke Rehabilitation Research, Kessler Foundation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMBarrett2
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Vascular Dementia; Memory Deficits
Keywords: Aricept; Donepezil; Memory; vascular dementia; stroke; functional tasks; self-generation
MeSH Terms: conditions — Stroke; Dementia, Vascular; Memory Disorders | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aricept- A (Experimental): Half of subjects are randomized to immediate treatment with donepezil 5mg orally daily following baseline testing, with retesting at 12 and 24 weeks.
  Interventions: Drug: Donepezil and self-generated memory training; Drug: Donepezil and experimenter-administered memory training
- A2-12-week waiting period (Experimental): The remaining nine subjects are randomized to testing followed by a 12-week waiting period. After the 12 week wait, this group of subjects is retested and begins taking donepezil, 5 mg orally daily, with retesting at 24 weeks
  Interventions: Drug: Donepezil and self-generated memory training; Drug: Donepezil and experimenter-administered memory training

INTERVENTIONS:
Drug: Donepezil and self-generated memory training — Aricept 5 mg PO qd for 4 weeks followed by Aricept 10 mg PO qd for 8 weeks
  Other Names: Aricept
Drug: Donepezil and experimenter-administered memory training — Aricept 5 mg PO daily for 4 weeks followed by Aricept 10 mg PO qd for 8 weeks
  Other Names: Aricept

SUMMARY:
Medications for memory improvement are available but they may not actually improve the ability to do real world tasks. The purpose of this research study is to determine if a medicine used to treat memory problems donepezil(Aricept) enhances the ability to remember steps of functional tasks and the actual ability to perform tasks relevant to real-life independence. Aricept is an FDA approved medication for the treatment of Alzheimer's disease. Aricept is an investigational drug for the purposes of this study, and is not approved for this purpose.

DETAILED DESCRIPTION:
All participants will receive a behavioral intervention as part of the testing protocol: they will be asked to generate words to complete a phrase as they read written steps to perform functional tasks. Mood will be assessed using the Geriatric Depression Scale.(see page 8) Participants will be asked to estimate their memory, immediate attention mood, functional tasks (performing cooking and financial task) and "ability to take medications correctly" (pre-test or "offline" ratings, abstract judgments of their own ability not based directly on performance). They will perform self-assessments of their cognitive, functional abilities and mood using Likert scales. They will mark each of 5 vertical (23.5 cm) lines centered on white paper to indicate their ability. Each line will be labeled for each domain.

To estimate of naming ability, show the subject the Likert Scale (attached) for the naming domain. Then explain: "This scale is to measure how well you think your ability to name. Here is the top where you will mark if you think your performance is perfect, here is the bottom if you think you are terrible. You may be somewhere in between. (broadly indicated the whole middle area) mark where you think your performance would belong on this scale".

This standard protocol will be used by the examiner in this study to explain each domain with specific types of tasks, and give subjects practical hypothetical examples of good and poor performance.

Ability to take medication: Functional memory as applied to medication compliance will be assessed with the Hopkins Medication Schedule (HMS). This test has two part, HMS and pill box. The test will serve as a good evaluation of subject's functional memory, which we suspect it will be most strongly affected by Anosognosia.

The HMS: the participant was read (and read along with) a hypothetical scenario in which her physician gave her 1 prescription for an antibiotic and for aspirin to treat an infection along with directions for taking each. The participant was then asked to plan a schedule for taking these medications and water during the course of a day, following the instructions provided.

ELIGIBILITY:
Inclusion Criteria:

1. I am 18 to100 yrs old.
2. I had one stroke 4 months to 5 yrs ago
3. I am not taking Aricept or other cholinesterase inhibitors (e.g. Exelon, Razadyne) or memantine (Namenda).

Exclusion Criteria:

1. I have history of dementia and or have been diagnosed with a memory disorder prior to my stroke.
2. I have been on anti-depressants or other cognitive enhancing drugs for less than 3 months and the dose is not stabilized yet.
3. I consume alcohol more than or equivalent of 4 ounces hard liquor weekly.
4. I am taking oral anticholinergic medications like Bethanechol, Bentyl or Detrol.
5. I am a woman of childbearing potential or I am pregnant or a nursing mother.
6. I have a history of chronic vomiting or diarrhea.
7. I am allergic to Aricept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-05; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Primary: To examine whether taking Aricept results in improvement at remembering steps of functional tasks. | 12 weeks

SECONDARY OUTCOMES:
To examine whether taking Aricept and actually performing functional tasks improves memory over that provided by a self-generation strategy. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A. M. Barrett, MD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

REFERENCES:
- [Background] Goverover Y, Chiaravalloti N, DeLuca J. The relationship between self-awareness of neurobehavioral symptoms, cognitive functioning, and emotional symptoms in multiple sclerosis. Mult Scler. 2005 Apr;11(2):203-12. doi: 10.1191/1352458505ms1153oa. PMID 15794396
- See also: Stroke page on Kessler Foundation website — https://kesslerfoundation.org/researchcenter/stroke/index.php